CLINICAL TRIAL: NCT05697354
Title: Harmonization and Application of Cognitive Rehabilitation Protocols Using New Technologies of Virtual Reality and Telemedicine, in Alzheimer's Disease
Brief Title: New Virtual Reality Technologies and Telemedicine for Cognitive Rehabilitation in Alzheimer's Disease
Acronym: TaskCog-IVN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Federica Alemanno, Psy.D., Ph.D., Responsible of the Neuropsychology Service, IRCCS San Raffaele Scientific Institute, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TaskCog-IVN
Record Dates: First submitted 2023-01-12; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet group (Experimental): The Tablet group will carry out the exercises using the Khymeia VRRS Home Tablet.
  Interventions: Procedure: Cognitive rehabilitation using interactive tablet
- App group (Experimental): The App group will perform the exercises on their smartphone using the Khymeia Medico Amico App.
  Interventions: Procedure: Cognitive rehabilitation using smartphone App Medico Amico

INTERVENTIONS:
Procedure: Cognitive rehabilitation using interactive tablet — the cognitive rehabilitation exercises will be administered using the Khymeia VRRS Home Tablet. Patients will be asked to actively carry out exercises focused on the following cognitive functions: language, attention, executive functions, verbal memory, visuo-spatial memory.
  Arms: Tablet group
Procedure: Cognitive rehabilitation using smartphone App Medico Amico — the cognitive rehabilitation exercises will be administered through patients' smartphone using the Medico Amico App. Patients will be asked to observe and concentrate on exercises focused on the following cognitive functions: language, attention, executive functions, verbal memory, visuo-spatial memory.
  Arms: App group

SUMMARY:
Main objective: To verify the effectiveness of a cognitive rehabilitation program in Alzheimer patients, based on virtual reality, delivered remotely, at the patient's home, with two distinct methods: a tablet or an App (on the patient's smartphone).

Total treatment duration: 2 months.

Main endpoint: Post rehabilitation assessment of the patient's cognitive level; Secondary endpoints: assessment of patients' quality of life quality of life and patients' and caregivers' satisfaction.

The neuropsychological assessment of the patients includes: Mini Mental State Examination (primary outcome), quality of life in Alzheimer's disease (QoL-AD), Geriatric Depression Scale (GDS). The following questionnaires will be submitted to caregivers: Beck Depression Inventory-II (BDI), System Usability Scale (SUS).

DETAILED DESCRIPTION:
Multicentric study involving the following 14 italian hospitals: San Raffaele Hospital of Milan, Fondazione Istituto Neurologico Carlo Besta, Istituto delle Scienze Neurologiche di Bologna, Fondazione Ca' Granda - Ospedale Maggiore Policlinico, Fondazione Don Carlo Gnocchi Onlus, Istituto Auxologico Italiano, Humanitas Mirasole, Istituti Clinici Scientifici Maugeri, Fondazione Istituto Neurologico Nazionale C. Mondino, Istituto Centro San Giovanni di Dio Fatebenefratelli, Fondazione Ospedale San Camillo, Fondazione Santa Lucia, Fondazione Policlinico Universitario Agostino Gemelli, Associazione Oasi Maria SS Onlus.

40 patients affected by Alzheimer's disease, with initial to severe cognitive impairment (MMSE 13-24), and 1 of their caregivers (total caregivers: N=40) will be included in the study (total n= 80 subjects).

The protocol provides for two treatment groups:

* Tablet group (total number = 20 patients): cognitive rehabilitation carried out in telemedicine at home with tablets (using Khymeia VRRS Home Tablet equipment).
* App group (total number = 20 patients): cognitive rehabilitation carried out in telemedicine at home with the App (Khymeia App Medico Amico).

Each AD patient, regardless of the severity of the cognitive impairment in progress, will be assigned to a treatment group. Allocation to the treatment group will be randomized by stratified randomization by severity of cognitive impairment (initial and moderate level, having MMSE between 24 and 18, vs., medium-severe level, having MMSE between 17 and 13).

Cognitive rehabilitation, for each group, will last two months. Patients will undergo 45 minutes of telehealth cognitive rehabilitation per day, 5 days a week, for a total duration of 2 months.

In both groups (Tablet or App), the rehabilitation exercises will be focused on the following cognitive functions:

* Language
* Attention
* Executive functions
* Verbal memory
* Visuo-spatial memory

Evaluations will be carried out PRE and POST treatment, remotely (patient and caregiver at home, neuropsychologist in hospital).

PRE Ratings:

* Within 7 days before the start of treatment;
* Patient assessments: Mini Mental State Examination (primary outcome), quality of life in Alzheimer's disease (QoL-AD), Geriatric Depression Scale (GDS);
* Caregiver assessments: Beck Depression Inventory-II (BDI).

POST Ratings:

* Within 7 days after the last treatment session;
* Patient assessments: Mini Mental State Examination (primary outcome), quality of life in Alzheimer's disease (QoL-AD), Geriatric Depression Scale (GDS);
* Caregiver assessments: Beck Depression Inventory-II (BDI), System Usability Scale (SUS).

Total study duration per participant: 2.5 months.

ELIGIBILITY:
Inclusion Criteria:

* inform consent
* Proven diagnosis of Alzheimer's disease;
* MMSE score between 13 and 24;
* Aged between 50 and 80 years;
* Stable drug therapy for at least 3 months.

Exclusion Criteria:

* Denial of informed consent;
* Psychiatric diseases;
* Relevant cerebrovascular damage;
* Disabling visual or hearing impairments;
* Psychosis;
* Major depression;
* Abuse of alcohol or drugs;
* Use of psychopharmacological agents that may interfere with test performance or treatment.
* Participation in study protocols with experimental drugs.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Change from Mini Mental State Examination after treatment | After 2 months of treatment
  Neuropsychological test for the evaluation of cognitive efficiency and the presence of cognitive impairment. The test consists of thirty items, which refer to seven different cognitive areas: orientation in time, orientation in space, memory, attention, and calculation, language, constructive ability. It ranges from 0 (poorest score) to 30 (normal cognition). An increase of the MMSE score indicate an improvement in general cognition.

SECONDARY OUTCOMES:
Change in Quality of life in Alzheimer's disease after treatment | After 2 months of treatment
  The QOL-AD is a 13-item questionnaire designed to investigate, through the patient and caregiver, the quality of life (QOL) of patients diagnosed with Alzheimer's disease (AD). It ranges from 13 to 52. An increase in the scores indicate an improvement of the quality of life.
Change in Geriatric Depression Scale after treatment | After 2 months of treatment
  Most widespread assessment scale for detecting depressive symptoms in frail elderly patients and in patients with dementia. It ranges from 0 (no depression) to 15 (probable depression). An increase in the GDS score indicates a worsening of the depression symptoms.
Change in Beck Depression Inventory-II after treatment | After 2 months of treatment
  The BDI is a self-report tool consisting of 21 items. It assesses common symptoms of depression, and is considered a valid and reliable tool for screening for depression in the general population. It ranges from 0 (no depression) to 63 (major depression). Higher scores indicate an increase in depression severity.
System Usability Scale after treatment | After 2 months of treatment
  The SUS is a Likert scale made up of ten elements which offers a global view of the subjective assessments of the usability of a system. Usability measurements consider several aspects: effectiveness (users can successfully achieve their goals), efficiency (how much effort and resources are spent to achieve those goals), and satisfaction (the experience was satisfactory). Scores range from 10 (poor satisfaction) to 100 (high satisfaction). High scores indicate a good satisfaction of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Alemanno, Psy.D, Ph.D., Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No